CLINICAL TRIAL: NCT02946112
Title: Relationship Between Shoulder Position and Neuromuscular Mechanosensitivity in Volleyball Players With Shoulder Pain
Brief Title: Shoulder Position in Volleyball Players With Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Collaborators: University of Alcala (Other)
Responsible Party: Principal Investigator, Fco. Javier Montanez Aguilera, Phd, Cardenal Herrera University
Other Study IDs: Cardenal Herrera CEU
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-10

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Shoulder pain: volleyball players with shoulder pain
- No shoulder pain: volleyball players without shoulder pain

SUMMARY:
The aim of this study is to assess the relationship between shoulder position and the presence of pain in volleyball players. To do this, will be measured pain sensation and the position of acromion process

DETAILED DESCRIPTION:
The position is defined as the alignment of body segments at a given time. The assessment of the position is part of the physical examination. Recent studies have shown that photometry can be a reliable method to assess posture. The measurement of angles can identify situations as the forward position of the head and shoulder protraction.

The aim of this study is to assess the position of the shoulder, using photometry by the measurement of angle between acromion process and seventh cervical vertebra, and the relationship with the presence of pain in volleyball players.

For this study will be recruited thirty nine volleyball players. The variables measured are pain sensation registered with a visual analog scale and the position of acromion process measurement with photometry

ELIGIBILITY:
Inclusion Criteria:

* over 16 years old
* minimum of 3 days per week of training
* with or without shoulder pain

Exclusion Criteria:

* less than 1 year practicing volleyball

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: volleyball players
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Photometry to measure shoulder position | Once, at baseline

SECONDARY OUTCOMES:
Visual analog scale to measure pain levels | Once, at baseline

CONTACTS AND LOCATIONS:
Overall Officials: F Javier Montañez-Aguilera, PhD, Study Chair — CEU Cardenal Herrera University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gangnet N, Pomero V, Dumas R, Skalli W, Vital JM. Variability of the spine and pelvis location with respect to the gravity line: a three-dimensional stereoradiographic study using a force platform. Surg Radiol Anat. 2003 Nov-Dec;25(5-6):424-33. doi: 10.1007/s00276-003-0154-6. Epub 2003 Sep 16. PMID 13680185
- [Result] Ruivo RM, Pezarat-Correia P, Carita AI. Intrarater and interrater reliability of photographic measurement of upper-body standing posture of adolescents. J Manipulative Physiol Ther. 2015 Jan;38(1):74-80. doi: 10.1016/j.jmpt.2014.10.009. Epub 2014 Nov 12. PMID 25467608
- [Result] Raine S, Twomey LT. Head and shoulder posture variations in 160 asymptomatic women and men. Arch Phys Med Rehabil. 1997 Nov;78(11):1215-23. doi: 10.1016/s0003-9993(97)90335-x. PMID 9365352
- [Result] Ozunlu N, Tekeli H, Baltaci G. Lateral scapular slide test and scapular mobility in volleyball players. J Athl Train. 2011 Jul-Aug;46(4):438-44. doi: 10.4085/1062-6050-46.4.438. PMID 21944077
- [Result] Koslow PA, Prosser LA, Strony GA, Suchecki SL, Mattingly GE. Specificity of the lateral scapular slide test in asymptomatic competitive athletes. J Orthop Sports Phys Ther. 2003 Jun;33(6):331-6. doi: 10.2519/jospt.2003.33.6.331. PMID 12839208
- [Result] Ribeiro A, Pascoal AG. Resting scapular posture in healthy overhead throwing athletes. Man Ther. 2013 Dec;18(6):547-50. doi: 10.1016/j.math.2013.05.010. Epub 2013 Jun 20. PMID 23791560
- [Result] Van Maanen CJ, Zonnenberg AJ, Elvers JW, Oostendorp RA. Intra/interrater reliability of measurements on body posture photographs. Cranio. 1996 Oct;14(4):326-31. doi: 10.1080/08869634.1996.11745985. PMID 9110628
- [Result] van Niekerk SM, Louw Q, Vaughan C, Grimmer-Somers K, Schreve K. Photographic measurement of upper-body sitting posture of high school students: a reliability and validity study. BMC Musculoskelet Disord. 2008 Aug 20;9:113. doi: 10.1186/1471-2474-9-113. PMID 18713477
- [Result] Griegel-Morris P, Larson K, Mueller-Klaus K, Oatis CA. Incidence of common postural abnormalities in the cervical, shoulder, and thoracic regions and their association with pain in two age groups of healthy subjects. Phys Ther. 1992 Jun;72(6):425-31. doi: 10.1093/ptj/72.6.425. PMID 1589462